CLINICAL TRIAL: NCT01511484
Title: You Are What You Eat: A Randomised Controlled Trial of an Appearance-based Dietary Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Perception Lab (Other)
Collaborators: Unilever R&D (Industry)
Responsible Party: Principal Investigator, David Perrett, Principal Investigator, University of St Andrews
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PerceptionLab001
Record Dates: First submitted 2011-12-23; First posted 2012-01-18 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Fruit and Vegetable Consumption
Keywords: fruit; vegetables; appearance; skin color; carotenoids; diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Information-only (Experimental): Selected pages from the British National Health Service (NHS) information booklets ["5 A Day, Just Eat More (fruit & veg)"; pages i, ii, 12-15, 20 & 21] and ["5 A Day, Just Eat More (fruit & veg): What's it all about?"; pages i-ii)] were provided to all participants on completion of baseline questionnaires. The pages provided information on recommended portion sizes, meal planning, health benefits and answered frequently asked diet-related questions
  Interventions: Behavioral: Information-only
- Generic-appearance intervention (Experimental): Participants in the generic appearance intervention group received images to illustrate the impact of fruit and vegetable consumption on skin appearance. Participants in this group were presented with gender congruent stimuli, constructed by averaging the facial shape and colour of four male/female faces.
  Participants viewed the gender-congruent set of the resulting stimuli in two forms. Firstly, after completion of baseline questionnaires, images were displayed on a computer monitor. Participants were instructed to select what they perceived as the healthiest face colour, which was recorded by the computer program over two trials.
  Participants in this group also received a take-home photo quality leaflet to further illustrate the effect of fruit and vegetable consumption on skin colour.
  Interventions: Behavioral: Generic appearance intervention
- Personalised appearance intervention (Experimental): Participants in this group received stimuli manipulated in identical ways to that received by the generic appearance-intervention group, except the illustrations were performed upon images of the participant's own face.
  Interventions: Behavioral: Personalised appearance intervention

INTERVENTIONS:
Behavioral: Information-only — Selected pages from the British National Health Service (NHS) information booklets ["5 A Day, Just Eat More (fruit & veg)"; pages i, ii, 12-15, 20 & 21] and ["5 A Day, Just Eat More (fruit & veg): What's it all about?"; pages i-ii)] were provided to all participants on completion of baseline questionnaires. The pages provided information on recommended portion sizes, meal planning, health benefits and answered frequently asked diet-related questions
  Arms: Information-only
Behavioral: Generic appearance intervention — Participants in the generic appearance intervention group received images to illustrate the impact of fruit and vegetable consumption on skin appearance. Participants in this group were presented with gender congruent stimuli, constructed by averaging the facial shape and colour of four male/female faces.
  Participants viewed the gender-congruent set of the resulting stimuli in two forms. Firstly, after completion of baseline questionnaires, images were displayed on a computer monitor. Participants were instructed to select what they perceived as the healthiest face colour, which was recorded by the computer program over two trials.
  Participants in this group also received a take-home photo quality leaflet to further illustrate the effect of fruit and vegetable consumption on skin colour.
  Arms: Generic-appearance intervention
Behavioral: Personalised appearance intervention — Participants in this group received stimuli manipulated in identical ways to that received by the generic appearance-intervention group, except the illustrations were performed upon images of the participant's own face.
  Arms: Personalised appearance intervention

SUMMARY:
This study investigated whether illustration of the facial appearance benefits of fruit and vegetable consumption is able to motivate increased intake of this food group. The investigators hypothesize that individuals witnessing illustrations of the impact of a healthy diet will exhibit improvements in diet relative to a control group receiving only information on the health-benefits of this food group.

ELIGIBILITY:
Inclusion Criteria:

* Student or staff member at University of St Andrews
* Has access to email account to receive link to weekly online questionnaire.

Exclusion Criteria:

* Exited study before completion
* Unable to make dietary changes due to a medical condition

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2011-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Fruit and vegetable consumption | up to 10 weeks
  Participants completed a computerised food frequency questionnaire to establish fruit and vegetable consumption. Participants were asked to retrospectively report consumption frequency of fruit juice, fruit, vegetable juice, salad, vegetable soup and vegetable items over the past seven days. Participants reported consumption of standard portion sizes and were provided with NHS illustrations of portion size guidelines to assist estimations.

CONTACTS AND LOCATIONS:
Overall Officials: Ross D Whitehead, MSc, Study Director — University of St Andrews
Locations (1):
- Perception Lab, School of Psychology, University of St Andrews, St Andrews, Fife, United Kingdom

REFERENCES:
- [Background] Stephen ID, Coetzee, V, Perrett D. Carotenoid and Melanin Pigment Coloration Affect Perceived Human Health. Evolution and Human Behaviour.32(3): 216-227. 2011.
- [Background] Stephen ID, Law Smith MJ, Stirrat MR, Perrett DI. Facial Skin Coloration Affects Perceived Health of Human Faces. Int J Primatol. 2009 Dec;30(6):845-857. doi: 10.1007/s10764-009-9380-z. Epub 2009 Oct 26. PMID 19946602
- [Background] Whitehead RD, Ozakinci G, Stephen ID, Perrett DI. Appealing to vanity: could potential appearance improvement motivate fruit and vegetable consumption? Am J Public Health. 2012 Feb;102(2):207-11. doi: 10.2105/AJPH.2011.300405. Epub 2011 Dec 15. PMID 22390433
- [Derived] Whitehead RD, Ozakinci G, Perrett DI. A randomized controlled trial of an appearance-based dietary intervention. Health Psychol. 2014 Jan;33(1):99-102. doi: 10.1037/a0032322. Epub 2013 Mar 25. PMID 23527517